CLINICAL TRIAL: NCT04909580
Title: Decision Coaching Using a Patient Decision Aid for Youth and Parents Considering Insulin Delivery Methods for Type 1 Diabetes: a Pretest Posttest Study
Brief Title: Decision Coaching for Youth and Parents Considering Insulin Delivery Methods for Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Margaret Lawson (Other)
Responsible Party: Sponsor-Investigator, Margaret Lawson, Pediatric Endocrinologist, Children's Hospital of Eastern Ontario
Organization: Children's Hospital of Eastern Ontario (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 11/76X
Record Dates: First submitted 2019-05-07; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Pre post study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- decision coaching (Experimental): Decision coaching with a patient decision aid guided by the Ottawa Decision Support Framework
  Interventions: Behavioral: Decision coaching with a patient decision aid

INTERVENTIONS:
Behavioral: Decision coaching with a patient decision aid — Decision coaching guided by the Ottawa Decision Support Framework

SUMMARY:
A pre-/post-test design. Youth with type 1 diabetes and their parent(s) were referred to the intervention by their diabetes physician. Decision coaching guided youth and their parents in completing a patient decision aid that was pre-populated with evidence on insulin delivery options. Primary outcomes were youth and parent scores on the low literary version of the Decisional Conflict Scale (DCS).

DETAILED DESCRIPTION:
A pre-/post-test design was used. Youth with type 1 diabetes and their parent(s) were referred to the intervention by their diabetes physician. Eligible participants were youth under 18 years old with T1D and their parents, who were considering a change in insulin delivery method, capable of participating in the decision making process, and able to read and speak English or French. No lower age limit was set for youth participants, provided the youth and parent(s) could participate in the consent or assent process. Family dyads (youth and one parent) and family triads (youth and two parents) were included.

The intervention was decision coaching guided by the Ottawa Decision Support Framework for youth with type 1 diabetes and their parents using a patient decision aid that was pre-populated with evidence on insulin delivery options.

ELIGIBILITY:
Inclusion Criteria:

* Youth with type 1 diabetes and their parents
* considering a change in their insulin delivery method
* capable of participating in the decision making process
* able to read and speak English or French

Exclusion Criteria:

* Using an insulin pump

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2013-09-05 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2015-12-05 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict | Change from baseline decision conflict scale 14 days after intervention
  Decision Conflict Scale - minimum score 0; maximum score 100

SECONDARY OUTCOMES:
Choice predisposition | Change from baseline predisposition scale to 14 days after intervention
  Choice Predisposition Scale - minimum score 0; maximum score 4
Preferred choice | Immediately after intervention
  Questionnaire asking participants for their preferred choice for insulin delivery method
Genetic Counselling Satisfaction Scale (modified version) | 14 days after the intervention
  Questionnaire that combined a shared decision making satisfaction rating tool and a modified version of the Genetic Counselling Satisfaction Scale

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L Lawson, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Lawson ML, Shephard AL, Feenstra B, Boland L, Sourial N, Stacey D. Decision coaching using a patient decision aid for youth and parents considering insulin delivery methods for type 1 diabetes: a pre/post study. BMC Pediatr. 2020 Jan 3;20(1):1. doi: 10.1186/s12887-019-1898-4. PMID 31900152